CLINICAL TRIAL: NCT00803543
Title: Seroprevalence of HSV-2 in HIV Infected Subjects and the Effect of Daiy Valacyclovir in the Reduction of HSV-2 Recurrences and Viral Shedding
Brief Title: Effect of Valacyclovir in the Reduction of HSV-2 Recurrence and Shedding
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Nicholas Van Wagoner, MD, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F080718009
Record Dates: First submitted 2008-12-03; First posted 2008-12-05 (Estimated); Results first posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-06

CONDITIONS: HIV; HIV Infections
Keywords: HSV-2; Herpes Simplex; HSV Type 2; HIV; HIV/HSV; treatment experienced
MeSH Terms: conditions — HIV Infections; Herpes Simplex | interventions — Valacyclovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Valacyclovir (Active Comparator): This is the arm taking Valacyclovir
  Interventions: Drug: Valacyclovir
- Placebo (Placebo Comparator): This is the arm taking the placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valacyclovir — 500 mg tablets. Dosage two tablets (1000 mg)once daily for 24 weeks
  Other Names: There are no other names
  Arms: Valacyclovir
Drug: Placebo — Dosage: Two tablets once a day for 24 weeks
  Other Names: There are no other names
  Arms: Placebo

SUMMARY:
The purpose of the study is to determine how common herpes is among persons with HIV who do not know they have it and if valacyclovir reduces outbreaks of herpes, the amount of HIV in the blood, and the amount of HSV in bodily secretions.

DETAILED DESCRIPTION:
Most people with herpes infections do not know they have the infection. HSV infections most often occur in areas in and around the mouth and genital tract. HSV Type 1 (HSV-1) usually causes "cold sores" or fever blisters and HSV Type 2 (HSV-2) usually causes lesions in the genital or rectal areas. However, HSV-1 can sometimes cause genital herpes and HSV-2 can cause oral lesions (acquired from oral-genital sex). Herpes Simplex is transmitted by contact with someone who is shedding virus in either the mouth or genital tract, usually by kissing or sexual intercourse. While contact with an active sore can cause transmission, so can contact with saliva or genital secretions that are infected, even when the person does not have an obvious sore. This is called asymptomatic shedding of HSV. Once acquired, the virus has the ability to remain inactive in the nervous system in the area of the mouth or genital region.

Persons with both HIV and HSV-2 often have shedding of both viruses. We know that persons with HSV-2 tend to have increased amounts of HIV in their blood as well. Recently, research studies have found that taking medicine daily to prevent asymptomatic HSV-2 shedding can reduce the amount of HIV found in the blood and in genital secretions. This study seeks to determine how common herpes is among persons with HIV who do not know they have it and if valacyclovir (FDA approved drug) reduces outbreaks of herpes, the amount of HIV in the blood, and the amount of HSV in bodily secretions.

ELIGIBILITY:
Inclusion Criteria:

* 19 years or older
* HSV-2 (Herpes simplex virus type 2) seropositive as determined by HerpeSelect-2 ELISA
* Documented HIV-1 seropositive
* Currently receiving HAART for 3 months or longer
* CD4 (cluster of differentiation 4) count 350 or greater
* Women of child bearing potential must agree to use acceptable contraceptive measures during the entire conduct of the study. Acceptable contraceptive methods include one or more of the following: oral hormonal contraceptives, injectable hormonal contraceptives, transdermal hormonal contraceptives, IUD (intrauterine device), diaphragm or cervical cap.
* Willing and able to provide written informed consent, undergo clinical evaluations, and take study drug as directed

Exclusion Criteria:

* History of symptomatic genital herpes, lesions or symptoms consistent with genital herpes, or recurrent undiagnosed symptoms consistent with genital herpes.
* Known history of adverse reaction to acyclovir, valacyclovir, or famciclovir.
* Planned open label use of acyclovir, valacyclovir, ganciclovir, valganciclovir, famciclovir, cidofovir, or foscarnet for oral herpes or other herpes viral infections.
* Medical history of seizures
* Renal insufficiency, defined as serum creatinine greater than 1.5 mg/dl
* AST (aspartate aminotransferase) or ALT (alanine aminotransferase) over 5 times uper limit of normal
* History of thrombotic microangiopathy
* For women, pregnancy as confirmed by a urine or serum pregnancy test.
* Any other condition which, in the opinion of the principal investigator, may compromise the subject's ability to follow study procedures and complete the study.
* Participants with active bacterial STDs (sexually transmitted diseases) may be treated and be eligible for enrollment 14 days after STD therapy is discontinued and symptoms have resolved.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2009-01; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Van Wagoner, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Community Care Building, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valacyclovir | Placebo
Started | 69 | 34
Completed | 45 | 22
Not Completed | 24 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valacyclovir | Placebo | Total
Number analyzed (Participants) | 45 | 22 | 67
Age, Continuous [Mean (Full Range); unit: years] | 45 [23 to 68] | 43 [27 to 61] | 45 [23 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 1 | 9
  Male | 37 | 21 | 58
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 45 | 22 | 67
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 25 | 9 | 34
  White | 20 | 13 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 45 | 22 | 67
Absolute CD4 (cluster of differentiation 4) Count [Mean (Full Range); unit: cell/ml] | 528 [165 to 1135] | 693 [198 to 1272] | 582 [165 to 1272]
Number with Undetectable Viral Load [Number; unit: participants] | 40 | 19 | 59

OUTCOME MEASURES:

1. Primary Outcome: Herpes Simplex Virus Type 2 Recurrence
Description: Number of recurrences of genital herpes
Time Frame: 24 Weeks
Population: No participants reported genital herpes recurrence during the study.
Measure: Number; unit: Recurrence
Arm/Group | Valacyclovir | Placebo
Number analyzed (Participants) | 45 | 22
Recurrence | 0 | 0

2. Primary Outcome: CD4 Count
Description: CD4 count as measured after 24 weeks of placebo versus valacyclovir. Reports as cells/ml
Time Frame: 24 weeks
Measure: Mean (Full Range); unit: cells/ml
Arm/Group | Valacyclovir | Placebo
Number analyzed (Participants) | 45 | 22
cells/ml | 536 [191 to 1112] | 627.5 [199 to 1268]

3. Primary Outcome: Number of Participants With an HIV Viral Load of <500 Copies/ml
Description: Number of participants with an HIV Viral Load of <500 copies/ml at 24 weeks
Time Frame: 24 weeks
Measure: Number; unit: Participants
Arm/Group | Valacyclovir | Placebo
Number analyzed (Participants) | 45 | 22
Participants | 38 | 20

4. Primary Outcome: Rate of Asymptomatic HSV-2 Genital Shedding
Description: Proportion of days on which HSV shedding was observed. This part of the study was performed in a subset of participants (N = 34). Participant collected daily genital specimens for 8 weeks starting at week 16 and continuing through week 24 of the study.
Time Frame: 24 weeks
Measure: Number; unit: Proportion of days
Units Other Than Participants: Total Number of Days Assessed
Arm/Group | Valacyclovir | Placebo
Number analyzed (Participants) | 26 | 8
Number analyzed (Total Number of Days Assessed) | 1456 | 448
Proportion of days | 0.0009 | 0.0001

ADVERSE EVENTS:
Time Frame: Entire study
Arm/Group | Valacyclovir | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/22
Other Adverse Events (participants affected / at risk) | 0/45 | 0/22

LIMITATIONS AND CAVEATS:
Small populations size. High level of patient withdrawal and loss to follow up.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No